CLINICAL TRIAL: NCT02265133
Title: Corneal Sensitivity and Nerve Fiber Morphology in Patients With Sleep Apnea Syndrome
Brief Title: Corneal Sensitivity in Patients With Sleep Apnea Syndrome
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Danielle Robertson, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU 102011-033
Record Dates: First submitted 2011-12-21; First posted 2014-10-15 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a prospective, single center clinical trial to assess corneal sensitivity and nerve fiber morphology in patients with sleep apnea compared to normal controls. Healthy volunteers with no history of ocular or uncontrollable systemic disease will be encouraged to participate in the study. After execution and review of the consenting procedures, a detailed history will be taken and a slit lamp examination performed, verifying ocular health. This consists of an examination of both eyes including assessments of ocular lids, lashes, cornea and conjunctival evaluation. Corneal touch thresholds will be tested with a Cochet-Bonnet aesthesiometer, a standard non-invasive measure of corneal sensitivity. Corneal nerves will be imaged using a modified HRT in vivo confocal microscope. The in vivo confocal microscope allows for high resolution imaging of the nerve plexus under the corneal epithelium. This corneal nerve plexus is responsible for corneal sensitively and changes or loss have been established as an early, sensitive indicator of corneal neuropathy. The investigators anticipate that this study will require approximately 30 patients for each group and will last approximately 12 months for recruitment and completion of subject visit phases. There is only one clinical visit designed for this project, unscheduled visits may be scheduled in case of an adverse event.

Patient recruitment will be complete at the one-year time point. At the 14 month time point, all data points will have been collected and assessment of the outcome measure (corneal sensitivity in sleep apnea patients versus control patients) will be complete.

DETAILED DESCRIPTION:
Screening Assessment: Following the execution of informed consent, subjects will be carefully screened for ocular signs and symptoms, consistent with the protocol inclusion and exclusion criteria. This includes review of ocular and medical history including use of concomitant & ocular medications and surgeries performed in the past. Researchers will also collect age, ethnicity, demographics, ophthalmic notes and eye exam history. Upon completion of the screening exam, subjects will be deemed eligible based on study criteria the testing procedures will be performed by the investigators.

Testing procedures: The visit will include:

Slit Lamp Microscopy:

An ocular examination of the external (lids, lashes) along with internal (cornea, lens, retina) structures of the eye can be performed with the aid of a slit lamp. This instruments uses lenses and an external light source that can be refracted at different angles and intensities to assess ocular structures for diagnostic purposes.

Corneal sensitivity measurement:

1. Corneal touch sensitivity will be determined using a Cochet-Bonnet aesthesiometer mounted on a standard slit lamp biomicroscope. The Cochet-Bonnet aesthesiometer is routinely used for clinical research purposes to investigate corneal touch thresholds.
2. For sensitivity measurements, a 0.12 mm diameter nylon thread will be slowly brought forward to briefly touch the cornea perpendicularly and then quickly withdrawn.
3. On each occasion, the patient will be asked to respond whenever a stimulus is felt.
4. Thread length is used to quantitatively assess sensitivity. The longest thread length is used first (6 cm), as this provides the lowest stimulus intensity.
5. If the subject is unable to detect the touch stimulus, the thread will be systematically shortened in length by 0.5 cm steps until the stimulus is felt.
6. The criterion for the sensitivity threshold will be the filament length which gives a 50% positive response from four stimulus applications.

In Vivo Confocal Microscope

1. Corneal nerves will be imaged using a modified in vivo confocal microscope which is routinely used in our clinics (HRT Rostock corneal module, Heidelberg Engineering).
2. The HRT In Vivo Confocal microscope was modified by adding a motor to automate the focus. This does not alter the integrity, the application, the intent or the light source of the instrument.
3. Corneas will be anesthetized with a topical anesthetic, proparacaine, prior to scanning.
4. The confocal microscope will briefly touch the patient's eye and the images saved for further analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking volunteers.
2. Patients with a diagnosis of sleep apnea.
3. Non-contact lens wearers of any gender and race, ages 18 and up.
4. Minority representation will be proactively encouraged.
5. Patients that are willing to review, understand, and sign the written Informed Consent.
6. Written authorization for use or release of health and research study information.
7. Patients that are willing and able to cooperate with the Investigator and follow all instructions.

Exclusion Criteria:

1. Use of ocular drops including over the counter (OTC) dry eye drops.
2. Previous history of corneal surgery.
3. Previous history of ocular trauma.
4. History of Diabetes Mellitus.
5. Current active or previous history of Herpes virus keratitis.
6. Current or former Contact lens wear.
7. Chronic history of dry eye disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sleep Apnea and normal controls
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Corneal Sensitivity | 1-Day
  To investigate whether diminished corneal sensitivity contributes to corneal problems commonly reported in patients with sleep apnea. Specifically, this study will correlate changes in corneal touch thresholds with corneal nerve fiber morphology using in vivo confocal microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Robertson, O.D, PhD, Principal Investigator — UTSW Medical Center at Dallas
Locations (2):
- United States (2):
  - Parkland Hospital, Dallas, Texas
  - Aston Ambulatory Care Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No